CLINICAL TRIAL: NCT02485678
Title: A Pragmatic Cluster-Randomized Trial of Ambulatory Toxicity Management in Patients Receiving Adjuvant or Neo-adjuvant Chemotherapy for Early Stage Breast Cancer (AToM)
Brief Title: A Pragmatic Trial of Ambulatory Toxicity Management in Patients Receiving Adjuvant or Neo-adjuvant Chemotherapy for Early Stage Breast Cancer
Acronym: AToM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: University Health Network, Toronto (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OCOG-2015-ATOM
Record Dates: First submitted 2015-06-10; First posted 2015-06-30 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Early Stage Breast Cancer
Keywords: ambulatory toxicity management; adjuvant or neoadjuvant chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proactive Telephone Toxicity Management (Experimental): Proactive Telephone Toxicity Management
  Interventions: Other: Proactive Telephone Toxicity Management; Other: PRO Sub-Study
- Control Arm (Active Comparator): Control
  Interventions: Other: Control Arm; Other: PRO Sub-Study

INTERVENTIONS:
Other: Proactive Telephone Toxicity Management — Centres randomized to this arm will implement a pro-active telephone toxicity management program, for all eligible early stage breast cancer patients beginning neo-adjuvant or adjuvant chemotherapy within the intervention period until the end of their systemic treatment. Patients will receive a phone call from a local nurse who has been trained on the toxicity management toolkit at 24-72 hours and at 8 to 10 days following each chemotherapy administration. The provider conducting the call will be provided with a script and will complete the Telephone Follow-Up Questionnaire which includes questions from the abbreviated NCI PRO-CTCAE tool. The nurse conducting the call will also be provided with the provider version of the symptom management booklet and provide toxicity management counseling. If any toxicity-related problems are identified during the call, a second call will take place 24 hours after the initial call to ensure the problem is resolving or to provide additional support.
  Arms: Proactive Telephone Toxicity Management
Other: Control Arm — Centres randomized to the control arm will continue to provide routine care for chemotherapy-related toxicities as is the current standard in the centre.
  Arms: Control Arm
Other: PRO Sub-Study — A sub-set of approximately 25 patients enrolled at each participating centre will participate in a Patient Reported Outcomes (PRO) sub-study to assess the effect of the intervention on secondary outcomes.

SUMMARY:
Comparison of the number of ER plus hospital visits that occurred during chemotherapy between the telephone intervention and control arms.

DETAILED DESCRIPTION:
Using a pragmatic cluster-randomized trial design, 20 Ontario cancer centres that provide care to patients with breast cancer will be randomly allocated to one of two arms: pro-active telephone toxicity management (intervention), or control (routine care). All patients with early stage (I-III) breast cancer who commence adjuvant or neo-adjuvant chemotherapy at participating institutions during the 6 to 12-month intervention period (will vary between centres depending on the number of incident cases) will be evaluated using Ontario healthcare administrative data. A sub-set of at least 25 patients at each participating institution will participate in a PRO sub-study involving the completion of standardized questionnaires to measure: a) severity of chemotherapy treatment toxicities; b) self-care for management of chemotherapy toxicities; c) self-efficacy (confidence) for managing symptoms; d) quality of life; and e) coordination of care. Patients participating in the PRO sub-study will be asked to provide consent to link their PRO data to Ontario healthcare administrative data so that correlations between the symptom self-assessments and Quality of Life (QoL) measures can be made with the administrative data on ED+H visits and use of supportive care medications. the investigators will compare the use of supportive care medications (i.e. anti-emetics, growth factors) by patients in the intervention and control arms to assess their influence on severity of chemotherapy-related toxicities as part of an exploratory sub-group analysis in patients >65 years of age as administrative data on supportive care medication use is only available for this age group.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Diagnosis of early stage (I-III) breast cancer
* Starting adjuvant or neo-adjuvant chemotherapy within the intervention period at a participating centre

Exclusion Criteria:

* Currently participating in a clinical trial involving an investigational agent

Inclusion Criteria for PRO Sub-Study

* Willingness to participate in the study and complete PRO questionnaires as required
* Ability to understand and provide written informed consent
* Language and literacy skills consistent with completing study questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Emergency and Hospital (ED+H) visits during chemotherapy | During chemotherapy and the 30 days post-chemotherapy
  Collect the number of ED+H visits that occurred during chemotherapy for all patients

SECONDARY OUTCOMES:
Severity of Chemotherapy | Assessed at baseline, at day 1 of cycle 2 prior to start of chemotherapy and again within 60 days of the completion of chemotherapy treatment
  Severity of treatment side effects will be measured using the NCI PRO CTCAE self-report tool (assessment on a 5 point scale).
Quality of Life (QOL) | Assessed at baseline, at day 1 of cycle 2 prior to start of chemotherapy and again within 60 days of the completion of chemotherapy treatment
  Measured using the Self-Care during Chemotherapy (L-PaSC), Stanford Self-Management Self-Efficacy Scale, FACT-B, GAD-7, PHQ-9, EQ-5D-3L
Coordination of Care | Assessed at baseline, at day 1 of cycle 2 prior to start of chemotherapy and again within 60 days of the completion of chemotherapy treatment
  Measured using the adapted Picker survey.
Health Economics | Initiation of chemotherapy to the end of chemotherapy plus 30 days
  Health system resources utilized by women receiving adjuvant or neo-adjuvant chemotherapy will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Monika Krzyzanowska, MD, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (20):
- Canada (20):
  - Royal Victoria Hospital, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Markham Stouffville, Markham, Ontario
  - Trillium Health Partners - The Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Cancer Centre, Newmarket, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre, Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Rouge Valley Health System, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Trillium Health Partners - Queensway Health Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario

REFERENCES:
- [Derived] Krzyzanowska MK, Julian JA, Gu CS, Powis M, Li Q, Enright K, Howell D, Earle CC, Gandhi S, Rask S, Brezden-Masley C, Dent S, Hajra L, Freeman O, Spadafora S, Hamm C, Califaretti N, Trudeau M, Levine MN, Amir E, Bordeleau L, Chiarotto JA, Elser C, Husain J, Laferriere N, Rahim Y, Robinson AG, Vandenberg T, Grunfeld E. Remote, proactive, telephone based management of toxicity in outpatients during adjuvant or neoadjuvant chemotherapy for early stage breast cancer: pragmatic, cluster randomised trial. BMJ. 2021 Dec 8;375:e066588. doi: 10.1136/bmj-2021-066588. PMID 34880055
- [Derived] Krzyzanowska MK, Julian JA, Powis M, Howell D, Earle CC, Enright KA, Mittmann N, Trudeau ME, Grunfeld E. Ambulatory Toxicity Management (AToM) in patients receiving adjuvant or neo-adjuvant chemotherapy for early stage breast cancer - a pragmatic cluster randomized trial protocol. BMC Cancer. 2019 Sep 5;19(1):884. doi: 10.1186/s12885-019-6099-x. PMID 31488084